CLINICAL TRIAL: NCT04444440
Title: Prophylactic Antibiotics During Treatment of Idiopathic Overactive Bladder With Intradetrusor onabotulinumtoxinA for the Reduction of Postoperative UTI: a Randomized Blinded Placebo-controlled Trial
Brief Title: Antibiotic Prophylaxis for Bladder Botox
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Women and Children's Health Research Institute, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00101838
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Overactive Bladder; Postoperative Urinary Tract Infection
Keywords: prophylaxis
MeSH Terms: interventions — Ciprofloxacin

STUDY DESIGN:
Intervention Model Description: Patients will be randomized at a 1:1 allocation ratio to two parallel treatment arms - intervention versus placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Active Comparator): Ciprofloxacin 500 mg PO every 12 hrs for 3 days following the procedure
  Interventions: Drug: Ciprofloxacin
- Placebo Arm (Placebo Comparator): Placebo pill PO every 12 hrs for 3 days following the procedure
  Interventions: Other: Placebo Pill

INTERVENTIONS:
Drug: Ciprofloxacin — Fluoroquinolone antibiotic.
  Arms: Treatment Arm
Other: Placebo Pill — Placebo Pill
  Arms: Placebo Arm

SUMMARY:
Injection of Botox into the bladder is a common treatment for overactive bladder. Postoperative bladder infection is one of the more frequently reported complications of this procedure. Prophylactic antibiotics given at the time of bladder Botox for the reduction of postoperative bladder infection have not been well studied. The main goal of our study is to determine if prophylactic antibiotics at the time of bladder Botox injection for the treatment of overactive bladder in women reduces postoperative bladder infection. The investigators are proposing a study which will randomize participants into two groups - one receiving Ciprofloxacin and the other receiving placebo pills for three days following the procedure. The primary outcome evaluated will be the difference in postoperative bladder infection between the two groups. The investigators will also investigate differences in reported side effects between the two groups possibly related to antibiotic use. Follow-up will be over six weeks following the procedure.

DETAILED DESCRIPTION:
This study will be a single-centred, double-blinded, randomized, placebo-controlled trial. Recruitment will be undertaken at two Urogynecology/Urology sites associated with the University of Alberta in Edmonton, Alberta. Participants will be randomized to treatment or placebo arm with a 1:1 allocation ratio. Patients and surgeons will be blinded.

On the day of the procedure, a urine culture will be collected preoperatively to identify pre-existing bacteriuria. Technique and dose of Botox injection will be at the discretion of the operating physician. Trigone-sparing technique with injection of 100 to 200 units of Botox distributed across 10 to 20 sites is generally used at our centre.

Follow-up will occur over a six-week postoperative period. A questionnaire will be used at each follow-up encounter to screen patients for urinary tract infection symptoms, voiding dysfunction, and other adverse events potentially related to the prophylactic antibiotics. Urine cultures will be collected to confirm infection for patients developing postoperative symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic OAB diagnosed clinically who have failed medical management
* Female
* Age ≥ 18

Exclusion Criteria:

* Patients with neurogenic OAB (OAB with potential underlying neurologic cause - multiple sclerosis, spinal cord injury, Parkinson's disease, other)
* Contraindication to injection of Botox - hypersensitivity to any botulinum toxin preparation or to any of the components in the formulation, current urinary tract infection, symptomatic urinary retention or PVR > 200 mL, unwillingness or inability to initiate CIC post-treatment if required.
* Contraindication to oral Ciprofloxacin - hypersensitivity or allergy to Ciprofloxacin or other fluoroquinolone, concurrently taking Tizanidine or Agomelatine.14
* Active antibiotic therapy for any indication at the time of Botox injection - increased risk of adverse reaction with combining antibiotics, reduced risk of UTI with additional antibiotic.
* Male
* Age < 18
* Pregnant and/or breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2021-06-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Postoperative Urinary Tract Infection | 2 weeks following the procedure
  new or worsening symptoms (dysuria, hematuria, frequency, urgency, suprapubic/flank pain, fever) AND positive urine culture (>10^5 CFU/mL)

SECONDARY OUTCOMES:
Rate of Postoperative Urinary Tract Infection Rate | 1 and 6 weeks following the procedure
  new or worsening symptoms (dysuria, hematuria, frequency, urgency, suprapubic/flank pain, fever) AND positive urine culture (>10^5 CFU/mL)
Rate of Other Adverse Events | 1, 2 and 6 weeks following the procedure
  New onset of side effects possibly related to Ciprofloxacin (nausea/vomiting, headache, abdominal pain, constipation, diarrhea, other)

CONTACTS AND LOCATIONS:
Locations (1):
- Urogynecology Clinic - Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No